CLINICAL TRIAL: NCT01514383
Title: Evaluation of Octylseal as a Topical Surgical Skin Incision Adhesive in General Surgery: A Case Series
Brief Title: Octylseal Surgical Adhesive in General Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R11-009
Record Dates: First submitted 2012-01-12; First posted 2012-01-23 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Wounds
Keywords: wounds
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgical Adhesive (Experimental): The surgical adhesive (cyanoacrylate) will be used once to close the topical skin surgical incision created during surgical procedures.
  Interventions: Device: Cyanoacrylate (Octylseal )

INTERVENTIONS:
Device: Cyanoacrylate (Octylseal ) — surgical adhesive
  Other Names: cyanoacrylate

SUMMARY:
The purpose of this study is to evaluate how surgical adhesive is used.

DETAILED DESCRIPTION:
In this Case Series Study, clinician experience and subject outcomes will be recorded in the use of a topical skin adhesive (Octylseal) on the closure of skin incisions from General surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for use of a topical surgical skin adhesive

Exclusion Criteria:

* Subjects with know sensitivity to topical surgical tissue adhesive products or degrading products (cyanoacrylates or formaldehyde)
* Subjects with a history of keloid formation, hypotension, insulin dependent diabetes mellitus, blood/clotting disorders, peripheral vascular diseases or hypertrophy history
* Subjects who present with a contraindications for product usage as per labeling
* A wound with evidence of active infection or gangrene or wounds of decubitus etiology
* Mucosal surfaces or across mucocutaneous junctions or skin that might be exposed to bodily fluids or with dense natural hair
* Subjects with known hypersensitivity to cyanoacrylate or formaldehyde

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ed Drower, MS, Study Director — Medline Industries
Locations (2):
- United States (2):
  - Jersey City Medical Center, Jersey City, New Jersey
  - Wyckoff Hospital, New York, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Surgical Adhesive
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Octylseal
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years]
  Adult | 47.5 (17.5)
  Pediatric | 11.3 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Wound Length Closure
Description: Primary incision wound length treatment in adult and pediatric general surgery
Time Frame: During Surgery
Measure: Mean (Standard Deviation); unit: milimeters
Arm/Group | Wound Length Closure of Paticipants Treated With Octylseal
Number analyzed (Participants) | 34
milimeters
  Adult | 28.97 (24.68)
  Pediatric | 21.00 (10.98)

2. Secondary Outcome: Number of Participants With a Score of "0" (No Hurt) on the Pain Rating Scale
Description: Pain was assessed using the Wong-Baker FACES™ Pain Rating Scale, with 0 =No Hurt to 10=Hurts Worst
Time Frame: At Surgery
Population: All 34 participants
Measure: Count of Participants; unit: Participants
Groups:
- No Pain Reported: Wong-Baker FACES™ Pain Rating Scale Pain Rating Scale from 0-10, with 0 =No Hurt to 10=Hurts Worst
Arm/Group | No Pain Reported
Number analyzed (Participants) | 34
Participants | 34

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Octylseal
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 1/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octylseal (N=34)
Infection (Infections and infestations) | 1 (1) — Of 74 incisions/lacerations treated in 34 patients, there was one (1) documented report of a possible incisional infection (1.4%). The complication was deemed not related to octylseal™.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No